CLINICAL TRIAL: NCT05426447
Title: Reduced Dietary Protein, Performance and Health
Brief Title: Protein and Performance (PROPER) in Endurance Athletes
Acronym: PROPER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Bente Kiens, Professor of Exercise, Nutrition and Metabolism, D Sci, PhD, Principal Investigator, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PROPER
Record Dates: First submitted 2021-09-22; First posted 2022-06-22 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Diet, Healthy; Protein Deficiency
Keywords: Diet intervention; Endurance athletes; Endurance performance; Skeletal muscle protein synthesis; Protein intake; Health markers; Microbiome
MeSH Terms: conditions — Protein Deficiency

STUDY DESIGN:
Intervention Model Description: A pair-matched group, parallel design within each sex
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced protein diet (Experimental): A 6-week eucaloric dietary intervention of reduced protein intake (~1g protein/kg body mass). The diet will, hence, contain ~7E% protein, ~63E% carbohydrate, and ~29E% fat.
  Participants are free-living and receive all food pre-packed from the study kitchen. The energy provision will be set to match energy balance.
  Interventions: Other: Dietary intervention of reduced protein intake
- Normal protein diet (Active Comparator): A 6-week eucaloric dietary intervention of normal protein intake (~2g protein/kg body mass). The diet will, hence, contain ~16E% protein, ~53E% carbohydrate, and ~30E% fat.
  Participants are free-living and receive all food pre-packed from the study kitchen. The energy provision will be set to match energy balance.
  Interventions: Other: Dietary intervention of normal protein intake

INTERVENTIONS:
Other: Dietary intervention of reduced protein intake — 6-wk dietary intervention of reduced protein intake
  Arms: Reduced protein diet
Other: Dietary intervention of normal protein intake — 6-wk dietary intervention of normal protein intake
  Arms: Normal protein diet

SUMMARY:
The present study is a parallel group design with randomised allocation to either a 1) reduced protein diet (RP) or a 2) normal protein diet (NP). The two groups will be pair-matched based on habitual dietary protein intake, endurance training, endurance performance, and sex.

The aim of the study is to investigate the effects of reducing dietary protein (~1g protein/kg body mass) compared to an eucaloric normal protein diet (~2g protein/kg body mass) for 6 weeks in well-trained endurance athletes on endurance performance, body composition, skeletal muscle protein synthesis, and health-related outcomes.

The hypothesis is that endurance performance will maintain or even be improved in well-trained endurance athletes after a 6-week dietary intervention of an eucaloric, protein reduced diet compared to a normal protein rich diet.

DETAILED DESCRIPTION:
Design: The present study will include two phases: a 3-week run-in period, and a 6-week intervention of controlled diets containing either a reduced dietary protein (RP) or normal (habitual) protein (NP). The run-in period serves as a period for obtaining general activity data and habitual dietary and training habits in order to match the groups before entering the dietary intervention period.

Subjects and dietary goals: The study is aiming at including 20 male endurance athletes exercising ~15hrs+/week. The 20 males will be pair-matched based on habitual endurance training, habitual dietary protein intake, and endurance performance, and allocated in a randomised order to: 1) a reduced-protein diet (RP) or 2) a normal-protein diet (NP).

3-weeks run-in period: After a minimum of 7 days after written consent has been obtained, the run-in period will begin. Habitual endurance training volumes will be registered in an online platform (TrainingPeaks) and daily activity level will be monitored using an accelerometer (SENS) throughout the run-in and diet intervention period. "Heavy water" (D2O) will be ingested in a large bolus (3.5ml/kg LBM) upon beginning of the run-in period and plasma enrichments will be maintained throughout the study period by ingesting small daily boluses. This serves to determine skeletal muscle protein synthesis throughout the study.

6-weeks dietary intervention: The diets will be eucaloric and the estimated energy percentages for macronutrients will be as follows: RP - Protein ~7E%, Carbohydrate ~63E%, Fat ~29E%. NP - Protein ~16E%, Carbohydrate ~53E%, Fat ~30E%. Weekly urine and faeces samples will be collected during the run-in period and dietary intervention and the controlled diets will be supplied weekly for the participants.

Testing: Extensive endurance performance and metabolic testing will be performed prior to-, and during the intervention on weeks -1, 0 (Pre), 3 (Mid), and 6 (Post). The tests include: Body composition by DXA-scanning, resting metabolic rate by online respirometry using a Vyntus (Jaeger, PCX), venous blood-, and skeletal muscle biopsy sampling from m. Vastus Lateralis, a standardised breakfasts, endurance cycling on an electro-magnetically braked bike (Lode Excalibur) or running on a motorised treadmill (Woodway), and haemoglobin mass measuring using a modified version of the CO-rebreathing method.

The body mass will be kept unchanged during the 6-weeks dietary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Endurance athlete
* Exercising at least 10hrs per week
* Habitual dietary protein intake ~2g/kg body mass
* BMI<25

Exclusion Criteria:

* Food allergies that exclude the controlled diet
* Inconsistent endurance training load

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Endurance performance on a bike | From Pre (week0) to post (week6)
  Endurance performance defined as maximal aerobic power (Wmax) during incremental test to exhaustion on a bike measured as 1-minute mean power output (W)
Microbiome | Run-in (week-3 to week0) vs dietary intervention (week0 to week6)
  Diversity of bacterial strains in gut microbiome measured in feces samples

SECONDARY OUTCOMES:
Resting metabolic rate | Pre (week0) to mid (week3)
  Measured in an over-night fasted state via indirect calorimetry expressed in MJ/day
Resting metabolic rate | Pre (week0) to Post (week6)
  Measured in an over-night fasted state via indirect calorimetry expressed in MJ/day
Lean body mass | Run-in (week-3) to Pre (week0)
  Measured by dual-energy x-ray (DXA)-scanningg expressed in kg
Lean body mass | Pre (week0) to Post (week6)
  Measured by dual-energy x-ray (DXA)-scanning expressed in kg
Total fat mass | Pre (week0) to Post (week6)
  Measured by dual-energy x-ray (DXA)-scanning expressed in kg
Total fat mass | Pre (week0) to mid (week3)
  Measured by dual-energy x-ray (DXA)-scanning expressed in kg
Total fat mass | Run-in (week-3) to Pre (week0)
  Measured by dual-energy x-ray (DXA)-scanning expressed in kg
Power output at 4mmol/L blood lactate | Pre (week0) to mid (week3)
  Alterations in Power output at 4mmol/L blood lactate in response to diet
Power output at 4mmol/L blood lactate | Pre (week0) to Post (week6)
  Alterations in Power output at 4mmol/L blood lactate in response to diet
Fractional utilisation of maximal oxygen uptake at 4mmol/L blood lactate | Pre (week0) to mid (week3)
  Alterations in Fractional utilisation of maximal oxygen uptake at 4mmol/L blood lactate in response to diet
Fractional utilisation of maximal oxygen uptake at 4mmol/L blood lactate | Pre (week0) to Post (week6)
  Alterations in Fractional utilisation of maximal oxygen uptake at 4mmol/L blood lactate in response to diet
Maximal oxygen uptake VO2peak | Pre (week0) to mid (week3)
  Alterations in Maximal oxygen uptake VO2peak measured by an online VO2 apparatus
Maximal oxygen uptake VO2peak | Pre (week0) to Post (week6)
  Alterations in Maximal oxygen uptake VO2peak measured by an online VO2 apparatus
Peak power output on a 10-seconds sprint | Pre (week0) to mid (week3)
  Alterations in peak power output on a 10-seconds sprint in response to diet
Peak power output on a 10-seconds sprint | Pre (week0) to Post (week6)
  Alterations in peak power output on a 10-seconds sprint in response to diet
Mean power output on a 10-seconds sprint | Pre (week0) to mid (week3)
  Alterations in mean power output on a 10-seconds sprint in response to diet
Mean power output on a 10-seconds sprint | Pre (week0) to Post (week6)
  Alterations in mean power output on a 10-seconds sprint in response to diet
Gross efficiency on a bike | Pre (week0) to mid (week3)
  Gross efficiency expressed as % of external power compared to internal (metabolic) power
Gross work efficiency on a bike | Pre (week0) to Post (week6)
  Gross efficiency expressed as % of external power compared to internal (metabolic) power
15-minute time-trial power output on a bike | Pre (week0) to mid (week3)
  Alterations in 15-minute time-trial mean power output
15-minute time-trial power output on a bike | Pre (week0) to Post (week6)
  Alterations in 15-minute time-trial mean power output
Fractional utilisation of maximal oxygen uptake during 15-minute time-trial | Pre (week0) to mid (week3)
  Alterations in Fractional utilisation of maximal oxygen uptake during 15-minute time-trial
Fractional utilisation of maximal oxygen uptake during 15-minute time-trial | Pre (week0) to Post (week6)
  Alterations in Fractional utilisation of maximal oxygen uptake during 15-minute time-trial
Respiratory exchange ratio | Pre (week0) to Post (week6)
  respiratory exchange ratio (RER) during rest and exercise using indirect calorimetry
Respiratory exchange ratio | Pre (week0) to Mid (week3)
  respiratory exchange ratio (RER) during rest and exercise using indirect calorimetry
Training load | Run-in (week-3) vs dietary intervention (week0 to week6)
  Training load as quantified by Edward's Training Impulse based on heart rate zones
Energy intake | Run-in (week-3) vs dietary intervention (week0 to week6)
  Habitual energy intake registered by food diaries expressed in Mega Joules
Energy expenditure | Run-in (week-3) vs dietary intervention (week0 to week6)
  Energy expenditure is measured by combining resting metabolic rate and daily activity recording from accelerometer data and heart rate monitor
Blood lactate concentration | Run-in (week-3 to week0) vs dietary intervention (week0 to week6)
  Glucose lactate measured in fasted state on an ABL800
Blood glucose concentration | Run-in (week-3 to week0) vs dietary intervention (week0 to week6)
  Glucose concentration measured in fasted state on an ABL800
Blood amino acid concentration | Run-in (week-3 to week0) vs dietary intervention (week0 to week6)
  Amino acid concentration measured by ELISA
Plasma metabolomics | Run-in (week-3 to week0) vs dietary intervention (week0 to week6)
  Plasma metabolomics by chromatography-mass spectrometry
Skeletal muscle protein expression | Pre (week0) to mid (week3)
  Alterations in Skeletal muscle protein expression
Skeletal muscle protein expression | Pre (week0) to Post (week6)
  Alterations in Skeletal muscle protein expression
Haemoglobin mass expressed in grams | Pre (week0) to mid (week3)
  Haemoglobin mass measured via inhalation of carbon monoxide (CO) using the modified CO-rebreathing method
Haemoglobin mass expressed in grams | Pre (week0) to Post (week6)
  Haemoglobin mass measured via inhalation of carbon monoxide (CO) using the modified CO-rebreathing method
Blood volume in ml | Pre (week0) to Post (week6)
  Blood volume measured via inhalation of carbon monoxide (CO) using the modified CO-rebreathing method
Blood volume in ml | Pre (week0) to Mid (week3)
  Blood volume measured via inhalation of carbon monoxide (CO) using the modified CO-rebreathing method
Energy expenditure measured as energy intake to maintain body weight | Run-in (week-3 to week0) vs dietary intervention (week0 to week6)
  Daily energy intake during intervention measured in Mega Joules

CONTACTS AND LOCATIONS:
Overall Officials: Nicki W Almquist, Post Doc, Study Director — University of Copenhagen; Bente Kiens, Professor, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No